CLINICAL TRIAL: NCT04390880
Title: IMPACT OF 18F-DCFPyL PET/CT ON INITIAL AND SUBSEQUENT TREATMENT STRATEGIES OF PATIENTS WITH PROSTATE CANCER (PROSPYL)
Brief Title: 18F-DCFPyL PET/CT Impact on Treatment Strategies for Patients With Prostate Cancer
Acronym: PROSPYL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-099757
Record Dates: First submitted 2020-05-04; First posted 2020-05-18 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; PET/CT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PEt/CT arm (Experimental): Subjects receive a PET/CT scan.
  Interventions: Drug: 18F-DCFPyL

INTERVENTIONS:
Drug: 18F-DCFPyL — Study participants will receive intravenous administration of 18F-DCFPyL and undergo a PET/CT imaging study. Patients may be reenrolled in the study, if 18F-DCFPyL PET/CT is performed for subsequent management decision.

SUMMARY:
The main purpose of this phase II trial study is to determine whether a positron emission tomography (PET)/computed tomography (CT) scan using 18F-DCFPyL affects the clinical management plan in Veterans.

In this study, the management plan prior to and after 18F-DCFPyL PET/CT will be recorded by specific questionnaires and corresponding changes in management will be analyzed. The scan will be used to see how the disease has spread. Both the treatment strategies and probable disease outcomes as relevant to clinical endpoints will be assessed. This study is open to Veterans only.

ELIGIBILITY:
Inclusion Criteria:

* Participants who fulfill criteria for initial staging or restaging as outlined below:

  1. Initial treatment strategy decisions (initial staging)

     All participants with histologically proven prostate cancer or strong suspicion of prostate adenocarcinoma based on very high PSA levels (>50 ng/mL) who require an initial treatment/management decision who may be candidate for any of the following strategies:

     A) Surgery B) External radiation therapy (RT) C) Other focal therapies D) Systemic medical treatment E) Watchful waiting
  2. Assessment for Subsequent treatment strategy (restaging), any of the following:

A) Participants with biochemical recurrence who are potential candidates for any salvage treatment. Biochemical recurrence is defined by rising PSA after definitive therapy with prostatectomy or radiation therapy, as any of the following:

1. Post radical prostatectomy (RP): PSA equals to or greater than 0.2 ng/mL measured more than 6 weeks after RP
2. Post-radiation therapy : Nadir + greater than or equal to 2 ng/mL rise in PSA B) Participants with known prostate cancer who undergo restaging because of new symptoms C) Participants with known metastatic prostate cancer who undergo restaging because of rising PSA with negative or inconclusive conventional imaging D) Participants with known prostate cancer who are treated medically or with RLT in whom response to treatment is assessed

   * Capability to provide written informed consent
   * Able to remain still for duration of each imaging procedure (about 30 minutes) * Participants may be reenrolled in the study, if 18F-DCFPyL PET/CT is performed for subsequent management decision.

Exclusion Criteria:

* Less than 18 years-old at the time of radiotracer administration
* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.)
* Any additional medical condition, serious concurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance.
* Inability to provide written informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gholam Berenji, M.D., Principal Investigator — Attending Physiscian
Locations (1):
- VA Greater Los Angeles Healthcare System, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PET/CT Arm
Started | 239
Completed | 238
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Subject with biopsy proven prostate cancer.
Arm/Group | PET/CT Arm
Number analyzed (Participants) | 239
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 206
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 239
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 86
  White | 107
  More than one race | 4
  Unknown or Not Reported | 32
Region of Enrollment [Number; unit: participants]
  United States | 239

OUTCOME MEASURES:

1. Primary Outcome: PRIMARY OBJECTIVES: I. To Determine the Impact of 18F-DCFPyL PET/CT on Initial and Subsequent Treatment Strategies of Patients With Prostate Cancer.
Description: the percentage of patients whose management was changed after PSMA PET/CT
Time Frame: 6 months
Measure: Number; unit: Percent
Arm/Group | PET/CT Arm
Number analyzed (Participants) | 74
Percent | 66.2

ADVERSE EVENTS:
Time Frame: 2 hours
Arm/Group | PET/CT Arm
All-Cause Mortality (participants affected / at risk) | 0/239
Serious Adverse Events (participants affected / at risk) | 0/239
Other Adverse Events (participants affected / at risk) | 0/239

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT04390880/Prot_SAP_000.pdf